CLINICAL TRIAL: NCT07395921
Title: Effects of Resveratrol Supplementation on Inflammatory Biomarkers and Cardiometabolic Parameters in Community-dwelling Adults. (RESINCA-trial)
Brief Title: Resveratrol Effects on Inflammatory Biomarkers and Cardiometabolic Parameters.
Acronym: RESINCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Research and Innovation Viña Concha y Toro (Industry)
Collaborators: Universidad Católica del Maule (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ECA Resveratrol - FIC
Record Dates: First submitted 2026-01-16; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Inflammation Biomarkers; Cardiometabolic Health Indicators; Antioxidant Status, Inflammation; Antioxidant Capabilities; Inflammaging
Keywords: Resveratrol; inflammation; inflammaging; antioxidant; cardiometabolic health; nutritional intervention
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: This Clinical Trial will be carried out with 3 parallel arms.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RES 120 (Sham Comparator): This is the control group
  Interventions: Dietary Supplement: RES 120
- RES 250 (Experimental): This is the experimental group 1
  Interventions: Dietary Supplement: RES 250
- RES 500 (Experimental): This is the experimental group 2
  Interventions: Dietary Supplement: RES 500

INTERVENTIONS:
Dietary Supplement: RES 120 — This grape pomace bar have 120 mg of total polyphenols contents
  Other Names: Nuvaoxi
  Arms: RES 120
Dietary Supplement: RES 250 — This grape pomace bar is enriched with resveratrol until reach 250 mg of total polyphenols contents
  Other Names: Nuvaoxi 250
  Arms: RES 250
Dietary Supplement: RES 500 — This grape pomace bar is enriched with resveratrol until reach 500 mg of total polyphenols contents
  Other Names: Nuvaoxi 500
  Arms: RES 500

SUMMARY:
This study aims to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on inflammatory biomarkers and cardiometabolic parameters in community-dwelling adults

DETAILED DESCRIPTION:
Three groups will be studied: control group (RES 120), experimental group 1 (RES 250) and experimental group 2 (RES 500).

During 8 weeks the RES 120 group will received daily one grape pomace bars with 120 mg of total polyphenols contents (TPC), the RES 250 group will received daily one grape pomace bars enriched with resveratrol until reach 250 mg of TPC and the RES 500 group will received daily one grape pomace bars enriched with resveratrol until reach 500 mg of TPC.

Outcomes will be assessed at baseline and after 8 weeks.

At the end of the study, the groups that shows less o no effects will be invited to enjoy the bar showing to be more effective.

Primary outcomes are: Total plasma antioxidant capacity (TAC), ultra-sensitivity CRP, IL-6, TNF-alfa, plasma malondialdehyde and AGEs.

Secondary outcomes are: body weight, Body Mass Index (BMI), basal metabolic rate, fat mass, skeletal muscle mass, and waist-to-hip ratio. Handgrip strength, 30-second sit-to-stand test, and heart rate variability. Fasting insulin, fasting glucose, HOMA-IR. Lipid profile, liver profile, blood pressure.

All procedures will be performed at the clinical simulation center of the Faculty of Medicine of the Catholic University of Maule.

The sample size was estimated under the following criteria, using G*Power software (version 3.1):

Primary outcome: Total Plasma Antioxidant Capacity (TAC). Type of comparison: differences between parallel groups. Level of significance (α): 0.05 (bilateral). Stat (1 - β): 80%. Minimum expected difference (Δ): 0.25 TAC units. Standard deviation (σ): 0.30 TAC units. Balanced allocation between groups (1:1:1). The minimum sample size required is 23 participants per group, considering an estimated loss or dropout rate of 15-20%, the sample size was increased to 27- 30 participants per group.

ELIGIBILITY:
Inclusion Criteria:

* Comunnity-dwelling persons.
* Any ethnicity.
* With willingness to consume the bar daily during the intervention period.

Exclusion Criteria:

* Allergy/intolerance to ingredients in the bar.
* Pregnancy or breastfeeding.
* Use of antioxidant/polymeroid supplements in the last 4 weeks.
* Unstable chronic diseases (e.g., severe liver failure, advanced kidney failure, active cancer).
* Persons in treatments that strongly interfere with polyphenol metabolism (e.g., antibiotics, anti-inflammatories, corticosteroids, anti-allergy medication).
* Persons with metal prosthesis.
* Persons undergoing or waiting for metabolic bariatric surgery.
* Persons with scheduled digestive surgery within the next 8 weeks
* Persons in recent treatments for hypertension (less than 3 month).
* Participation in another clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Inflammatory biomarkers: Total plasma antioxidant capacity (µmol/L). | From enrollment to the end of treatment at 8 weeks
  The total plasma antioxidant capacity by Ferric Reducing Antioxidant Power will assess with a blood sample pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on inflammatory biomarkers in community-dwelling adults.
Inflammatory Biomarkers: Ultra-sensitivity CRP (mg/L). | From enrollment to the end of treatment at 8 weeks
  The ultra-sensitivity CRP by Elisa test will assess with a blood sample pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on inflammatory biomarkers in community-dwelling adults.
Inflammatory Biomarkers: IL-6 (pg/mL). | From enrollment to the end of treatment at 8 weeks
  The IL-6 by Elisa test will assess with a blood sample pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on inflammatory biomarkers in community-dwelling adults.
Inflammatory Biomarkers: Plasma malondialdehyde (µmol/L). | From enrollment to the end of treatment at 8 weeks
  The plasma malondialdehyde by TBARS/HPLC method will assess with a blood sample pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on inflammatory biomarkers in community-dwelling adults.
Inflammatory Biomarkers: TNF-alfa (pg/mL). | From enrollment to the end of treatment at 8 weeks
  The TNF-alfa by Elisa test will assess with a blood sample pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on inflammatory biomarkers in community-dwelling adults.
Inflammatory Biomarkers: Advanced glycation end-products (AGEs) in 1 to 5 units. | From enrollment to the end of treatment at 8 weeks
  The AGEs will assess with non-invasive fluorescence pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on inflammatory biomarkers in community-dwelling adults.

SECONDARY OUTCOMES:
Cardiometabolic Parameters: Body weight (kg). | From enrollment to the end of treatment at 8 weeks
  Body weight will assess with electrical bioimpedance pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on cardiometabolic parameters in community-dwelling adults.
Cardiometabolic Parameters: Body mass index-BMI (kg/m2). | From enrollment to the end of treatment at 8 weeks
  The BMI will assess with electrical bioimpedance pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on cardiometabolic parameters in community-dwelling adults.
Cardiometabolic Parameters: Basal metabolic rate (kcal). | From enrollment to the end of treatment at 8 weeks
  The basal metabolic rate will assess with electrical bioimpedance pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on cardiometabolic parameters in community-dwelling adults.
Cardiometabolic Parameters: Fat mass (kg, %). | From enrollment to the end of treatment at 8 weeks
  The fat mass will assess with electrical bioimpedance pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on cardiometabolic parameters in community-dwelling adults.
Cardiometabolic Parameters: Skeletal muscle mass (kg). | From enrollment to the end of treatment at 8 weeks
  The skeletal muscle mass will assess with electrical bioimpedance pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on cardiometabolic parameters in community-dwelling adults.
Cardiometabolic Parameters: Waist-to-hip ratio. | From enrollment to the end of treatment at 8 weeks
  The waist-to-hip ratio will assess with electrical bioimpedance pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on cardiometabolic parameters in community-dwelling adults.
Cardiometabolic Parameters: Handgrip strength (kg). | From enrollment to the end of treatment at 8 weeks
  The handgrip strength will assess with dynamometry pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on cardiometabolic parameters in community-dwelling adults.
Cardiometabolic Parameters: 30-second sit-to-stand test (n° of repetitions achieved). | From enrollment to the end of treatment at 8 weeks
  The 30-second sit-to-stand test will assess with a 43 cm height chair pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on cardiometabolic parameters in community-dwelling adults.
Cardiometabolic parameters: HRV, RMSSD and SDNN in (ms). | From enrollment to the end of treatment at 8 weeks
  The heart rate variability will assess in 10 minutes with continuous recording of the resting electrocardiographic tracing pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on cardiometabolic parameters in community-dwelling adults.
Cardiometabolic parameters: PNN50 (%). | From enrollment to the end of treatment at 8 weeks
  The heart rate variability will assess in 10 minutes with continuous recording of the resting electrocardiographic tracing pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on cardiometabolic parameters in community-dwelling adults.
Cardiometabolic parameters: Insuline (µIU/mL). | From enrollment to the end of treatment at 8 weeks
  The fasting insulin by immunoassay will assess by a blood sample pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on cardiometabolic parameters in community-dwelling adults.
Cardiometabolic parameters: Glucose (mg/dL). | From enrollment to the end of treatment at 8 weeks
  The fasting glucose by enzymatic method will assess by a blood sample pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on cardiometabolic parameters in community-dwelling adults.
Cardiometabolic parameters: HOMA-IR (index). | From enrollment to the end of treatment at 8 weeks
  The HOMA-IR (calculated by fasting glucose x fasting insulin/405) will assess by a blood sample pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on cardiometabolic parameters in community-dwelling adults.
Cardiometabolic parameters: Lipid profile (mg/dL). | From enrollment to the end of treatment at 8 weeks
  The lipid profile: total cholesterol, LDL, HDL and Triglycerides by enzymatic method will assess with a blood sample pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on cardiometabolic parameters in community-dwelling adults.
Cardiometabolic parameters: Liver profile (U/L). | From enrollment to the end of treatment at 8 weeks
  The liver profile: ALS, AST, GGT: by enzymatic method will assess with a blood sample pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on cardiometabolic parameters in community-dwelling adults.
Cardiometabolic parameters: Blood pressure (mmHg) | From enrollment to the end of treatment at 8 weeks
  The systolic and diastolic blood pressure will assess with a sphygmomanometer pre and post intervention to evaluate the effect of the supplementation of grape pomace bars enriched in resveratrol on cardiometabolic parameters in community-dwelling adults.

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Casaubon Cruzat, Study Director — Center for Research and Innovation Viña Concha y Toro
Locations (1):
- Universidad Católica del Maule, Talca, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: No
In order to protect the privacy, data will be stored and coded. At the end of the study, data may be available upon a reasonable request and ensuring the participants' data confidentiality will be preserved.

REFERENCES:
- [Background] Chiva-Blanch, G., & Badimon, L. (2017). Effects of Polyphenol Intake on Metabolic Syndrome: Current Evidences from Human Trials. Oxidative medicine and cellular longevity, 2017, 5812401. https://doi.org/10.1155/2017/5812401
- [Background] Breuss, J. M., Atanasov, A. G., & Uhrin, P. (2019). Resveratrol and Its Effects on the Vascular System. International journal of molecular sciences, 20(7), 1523. https://doi.org/10.3390/ijms20071523
- [Background] Huang, H., Chen, G., Liao, D., Zhu, Y., Pu, R., & Xue, X. (2016). The effects of resveratrol intervention on risk markers of cardiovascular health in overweight and obese subjects: a pooled analysis of randomized controlled trials. Obesity reviews : an official journal of the International Association for the Study of Obesity, 17(12), 1329-1340. https://doi.org/10.1111/obr.12458
- [Background] Springer, M., & Moco, S. (2019). Resveratrol and Its Human Metabolites-Effects on Metabolic Health and Obesity. Nutrients, 11(1), 143. https://doi.org/10.3390/nu11010143
- [Background] Pastor, R. F., Restani, P., Di Lorenzo, C., Orgiu, F., Teissedre, P. L., Stockley, C., Ruf, J. C., Quini, C. I., Garcìa Tejedor, N., Gargantini, R., Aruani, C., Prieto, S., Murgo, M., Videla, R., Penissi, A., & Iermoli, R. H. (2019). Resveratrol, human health and winemaking perspectives. Critical reviews in food science and nutrition, 59(8), 1237-1255. https://doi.org/10.1080/10408398.2017.1400517
- [Background] Chudzińska, M., Rogowicz, D., Wołowiec, Ł., Banach, J., Sielski, S., Bujak, R., Sinkiewicz, A., & Grześk, G. (2021). Resveratrol and cardiovascular system-the unfulfilled hopes. Irish journal of medical science, 190(3), 981-986. https://doi.org/10.1007/s11845-020-02441-x
- [Background] Hou, C. Y., Tain, Y. L., Yu, H. R., & Huang, L. T. (2019). The Effects of Resveratrol in the Treatment of Metabolic Syndrome. International journal of molecular sciences, 20(3), 535. https://doi.org/10.3390/ijms20030535
- [Background] Mousavi SM, Milajerdi A, Sheikhi A, Kord-Varkaneh H, Feinle-Bisset C, Larijani B, Esmaillzadeh A . Resveratrol supplementation significantly influences obesity measures: a systematic review and dose-response meta-analysis of randomized controlled trials. Obes Rev. 2019 Mar;20(3):487-498. doi: 10.1111/obr.12775. Epub 2018 Dec 05.